CLINICAL TRIAL: NCT06667310
Title: Evaluatıon Of The Effect Of Neutrophıl/Lymphocyte, Platelet/Lymphocyte, Crp/Albumın, Base Defıcıt And Lactate Levels On Mortalıty Durıng The Admıssıon Of Trauma Patıents To Intensıve Care
Brief Title: Effects of Neutrophil/Lymphocyte, Platelet/Lymphocyte, CRP/Albumin and Lactate on Mortality in Trauma Patients Admitted to Intensive Care
Status: Completed | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Veli Fahri Pehlivan, Assistant Professor, Harran University
Other Study IDs: Hasan
Record Dates: First submitted 2024-10-25; First posted 2024-10-31 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Intensive Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intensive care units are medical units where patients are closely monitored 24 hours a day due to critical health problems that threaten their lives and where rapid interventions are made when necessary. The clinical conditions of patients in these units can change rapidly. There are many studies in the literature indicating that inflammation indicators such as Neutrophil/Lymphocyte, Platelet/Lymphocyte and C-Reactive Protein/Albumin ratios and blood gas values such as Lactate and Base Deficit are simple, cheap and rapid biomarkers that can provide an early idea about the clinical course of patients.

DETAILED DESCRIPTION:
Intensive care units are medical units where patients are closely monitored 24 hours a day due to critical health problems that threaten their lives and where rapid interventions are made when necessary. The clinical conditions of patients in these units can change rapidly. There are many studies in the literature indicating that inflammation indicators such as Neutrophil/Lymphocyte, Platelet/Lymphocyte and C-Reactive Protein/Albumin ratios and blood gas values such as Lactate and Base Deficit are simple, cheap and rapid biomarkers that can provide an early idea about the clinical course of patients. The researchers aimed to evaluate the relationship between Neutrophil/Lymphocyte, Platelet/Lymphocyte and C-Reactive Protein/Albumin ratios and biomarkers such as Lactate and Base Deficit with the clinical course and survival of trauma patients admitted to the ICU and to see the compatibility of our data with the existing literature.

ELIGIBILITY:
Inclusion Criteria:

* 1. All trauma patients admitted to our general intensive care unit

Exclusion Criteria:

- 1. Patients whose follow-up and treatment started and completed in the services.

2. Patients whose data is missing or whose data cannot be accessed.

Ages: 1 Year to 95 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1-95 age intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Primary outcome | one day
  1. LACTATE LEVELS RATİO MEASUREMENT

SECONDARY OUTCOMES:
seconary outcome | one day
  The effect of these measurements on mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Veli Fahri Pehlivan, Karaköprü, Şanliurfa, Turkey (Türkiye)